CLINICAL TRIAL: NCT03087019
Title: A Phase II Trial of Pembrolizumab With or Without Radiation in Patients With Recurrent or Metastatic Adenoid Cystic Carcinoma
Brief Title: Pembrolizumab With or Without Radiation in Patients With Recurrent or Metastatic Adenoid Cystic Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Jonathan Schoenfeld, MD, MPH, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-609
Record Dates: First submitted 2017-03-13; First posted 2017-03-22 (Actual); Results first posted 2021-04-22 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Adenoid Cystic Carcinoma
Keywords: adenoid cystic carcinoma
MeSH Terms: conditions — Carcinoma, Adenoid Cystic | interventions — Radiation; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab + Radiation (Experimental): * Up to 5 metastatic lesions targeted with radiation
  * Over 5 fractions starting within 7 calendar days following the first dose of pembrolizumab
  * Pembrolizumab will be administered on day 1 of each 21day cycle
  * Pembrolizumab is delivered intravenously
  Interventions: Radiation: Radiation; Drug: Pembrolizumab
- Pembrolizumab (Experimental): * Pembrolizumab will be administered on day 1 of each 21day cycle
  * Pembrolizumab is delivered intravenously
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Radiation: Radiation — Standard use of radiation is administered
  Arms: Pembrolizumab + Radiation
Drug: Pembrolizumab — Pembrolizumab is designed to restore the natural ability of the immune system to recognize and target cancer cells.
  Other Names: Keytruda

SUMMARY:
This research study is studying immunotherapy with or without radiation therapy as a possible treatment for adenoid cystic carcinoma.

The immunotherapy involved in this study is:

* Pembrolizumab (MK-3475 or KEYTRUDA).

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational agent to learn whether it works in treating a specific disease. "Investigational" means that the drug is being studied.

Pembrolizumab (MK-3475 or KEYTRUDA) is a humanized monoclonal antibody. An antibody is a common type of protein made in the body in response to a foreign substance (particles not typically found in your body such as bacteria or viruses). Antibodies attack foreign substances and protect against infection. Antibodies can also be produced in the laboratory for use in treating patients. Pembrolizumab is designed to restore the natural ability of the immune system to recognize and target cancer cells.

The FDA recently granted approval to pembrolizumab as a treatment for patients with recurrent or metastatic head and neck squamous cell carcinoma. Pembrolizumab has not been approved for treatment against adenoid cystic carcinoma.

This study is testing whether pembrolizumab with or without radiation is useful for patients with adenoid cystic carcinoma. Radiation therapy may be used to treat some ACC tumors that have spread to other parts of the body or recurred after surgery. Radiation therapy may affect the immune system to improve the efficacy of pembrolizumab

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed adenoid cystic carcinoma with evidence of recurrent or metastatic disease not amenable to potentially curative surgery or radiotherapy.
* Participants must have at least two RECIST v1.1 measurable non-CNS based lesions. Palliative radiation must be indicated for at least one of these lesions, and this lesion must be a candidate for radiation to a dose of 30 Gy of radiation over 5 fractions as deemed by a treating radiation oncologist. Documentation of volume and prescription isodose line will be collected. Re-irradiation of a previously treated lesion is not allowed. One lesion must be in a location where it will not be incorporated into the radiation fields so systemic response can be assessed. However, inclusion of patients with more than 10 measurable lesions is strongly discouraged and all patients must have life expectancy > 6 months.
* Participants must agree to undergo a research biopsy, if tumor is safely accessible, at baseline and after 2 cycles of pembrolizumab. Participants can be exempt if archival tumor tissue has been collected within 12 months of study enrollment that the Principal Investigator deems it appropriate/sufficient for analysis on this protocol. Biopsy of a lesion outside of the potential radiation treatment field is preferred to maintain consistency across cohorts.
* Participants must have archival tissue from the primary tumor or metastases available for correlative studies. Either a paraffin block or twenty unstained slides are acceptable. If twenty slides are not available, a lesser amount may be acceptable after discussion with the Principal Investigator.
* Prior systemic therapy: At least 2 weeks must have elapsed since the end of prior chemotherapy, biological agents (4 weeks for anti-cancer monoclonal antibody containing regimens) or any investigational drug product, with adequate recovery of treatment-related toxicity to NCI CTCAE Version 4.0 grade ≤1 (or tolerable grade 2) or back to baseline (except for alopecia or neuropathy). Any number of prior therapies for recurrent/metastatic ACC are allowed, with the exception of previous treatment with PD-1 pathway inhibitors.
* Prior radiation therapy: At least 3 weeks must have elapsed from prior radiation therapy. The prior site of radiotherapy must be documented as reirradiation of the same site is not allowed in this protocol.
* Be ≥ 18 years of age on day of signing informed consent.
* Have a performance status of 0 or 1 on the ECOG Performance Scale (see Appendix A).
* Participants must have documentation of a new or progressive lesion on a radiologic imaging study performed within 12 months prior to study enrollment (progression of disease over any interval is allowed) and/or new/worsening disease related symptoms within 12 months prior to study enrollment. This assessment is performed by the treating investigator. Evidence of progression by RECIST criteria is not required.
* Demonstrate adequate organ function as defined in Table 1, all screening labs should be performed within 10 days of treatment initiation.

Table 1 Adequate Organ Function Laboratory Values System Laboratory Value

* Hematological

  * Absolute neutrophil count (ANC) ≥1,500 /mcL
  * Platelets ≥100,000 / mcL
  * Hemoglobin ≥9 g/dL or ≥5.6 mmol/L without transfusion or EPO dependency (within 7 days of assessment)
* Renal
* Serum creatinine OR Measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤1.5 X upper limit of normal (ULN) OR ≥60 mL/min for subject with creatinine levels > 1.5 X institutional ULN
* Hepatic

  * Serum total bilirubin ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN
  * AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN OR ≤ 5 X ULN for subjects with liver metastases
  * Albumin >2.5 mg/dL
* Coagulation

  * International Normalized Ratio (INR) or Prothrombin Time (PT)
  * Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Creatinine clearance should be calculated per institutional standard.
* Baseline tumor measurements must be documented from tests within 28 days of study entry. Other non-laboratory tests must be performed within 28 days of study entry.
* Female subjects of childbearing potential should have a negative urine or serum pregnancy within 7 days prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female and male subjects of childbearing potential must agree to use an adequate method of contraception, as outlined in section 5.6, prior to study entry, for the duration of study participation, and 4 months after completion of pembrolizumab administration. Contraception is required starting with the first dose of study medication through 120 days after the last dose of study medication.
* Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
* Be willing and able to provide written informed consent for the trial.

Exclusion Criteria:

* Metastatic disease impinging on the spinal cord or threatening spinal cord compression. Patients that have had previous treatment of disease with impinging on the cord with either surgery or radiotherapy with clinical or radiographic evidence of response or stability are eligible.
* Surgical fixation of bone lesion to be irradiated is required and indicated to provide mechanical stability.
* Participant has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment), have no evidence of new or enlarging brain metastases, and are not using steroids for the purposes of treating brain metastasis induced edema for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability, because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Prior treatment with PD-1 or PD-L1 inhibitor
* Concurrent administration of other cancer specific therapy or investigational agents during the course of this study is not allowed.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Has a known history of active TB (Bacillus Tuberculosis)
* History of allergic reactions or hypersensitivity to pembrolizumab or any of its excipients.
* Uncontrolled intercurrent illness including but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Has known history of, or any evidence of active, non-infectious pneumonitis.
* Has an active infection requiring systemic therapy.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Subjects who are pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment. Pregnant women are excluded from this study because immunotherapy has the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk of adverse events in nursing infants secondary to treatment of the mother with immunotherapy, breastfeeding should be discontinued if the mother is treated on this protocol. Women who could potentially become pregnant while undergoing treatment on this protocol must be willing to use 2 methods of contraception.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has received a live vaccine within 30 days of planned start of study therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-04-25 (Actual); Primary Completion 2020-08-04 (Actual); Study Completion 2020-08-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Schoenfeld, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mahmood U, Bang A, Chen YH, Mak RH, Lorch JH, Hanna GJ, Nishino M, Manuszak C, Thrash EM, Severgnini M, Sanborn M, Sridharan V, Margalit DN, Tishler RB, Busse PM, Willers H, Mamon HJ, Yoo HJ, Pai SI, Wirth LJ, Haddad RI, Chau NG, Schoenfeld JD. A Randomized Phase 2 Study of Pembrolizumab With or Without Radiation in Patients With Recurrent or Metastatic Adenoid Cystic Carcinoma. Int J Radiat Oncol Biol Phys. 2021 Jan 1;109(1):134-144. doi: 10.1016/j.ijrobp.2020.08.018. Epub 2020 Aug 8. PMID 32781104

RESULTS

PARTICIPANT FLOW:
Groups:
- Pembrolizumab + Radiation: * Up to 5 metastatic lesions targeted with radiation
  * Over 5 fractions starting within 7 calendar days following the first dose of pembrolizumab
  * Pembrolizumab will be administered on day 1 of each 21day cycle
  * Pembrolizumab is delivered intravenously
  Radiation: Standard use of radiation is administered
  Pembrolizumab: Pembrolizumab is designed to restore the natural ability of the immune system to recognize and target cancer cells.
- Pembrolizumab: * Pembrolizumab will be administered on day 1 of each 21day cycle
  * Pembrolizumab is delivered intravenously
  Pembrolizumab: Pembrolizumab is designed to restore the natural ability of the immune system to recognize and target cancer cells.
Period: Overall Study
Arm/Group | Pembrolizumab + Radiation | Pembrolizumab
Started | 11 | 10
Completed | 10 | 10
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab + Radiation | Pembrolizumab | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 7 | 12
  >=65 years | 6 | 3 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 4 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 9 | 9 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Patients Demonstrating Objective Response In Non-Irradiated Lesions (Tumor Size on Scans)
Description: Objective response will be assessed in non-irradiated lesions among all eligible and treated patients pursuing RECIST 1.1. Per RECIST guidelines for target lesions, Complete Response (CR): disappearance of all target lesions; Partial Response (PR): >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD): >20% increase in sum of the longest diameter (LD) of measured lesions, referencing the smallest sum LD, or new lesions; Stable Disease (SD): neither PR nor PD. Objective response refers to tumor shrinkage at least qualifying as PR.
Time Frame: 2 years
Population: 21 subjects were enrolled. One subject withdrew consent before starting treatment and was replaced. A total of 20 patients (10 per each arm) received protocol treatment. Among 20 patients treated, 1 patient withdrew consent in order to pursue hospice care after receiving a single dose of pembrolizumab and was not evaluable for response.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Radiation | Pembrolizumab
Number analyzed (Participants) | 10 | 9
Participants | 0 | 0

2. Secondary Outcome: Progression Free Survival (Time From Randomization to Disease Progression or Death)
Description: Progression-free survival is defined as the time from randomization to disease progression or death, whichever occurs first. Patients who are alive without disease progression will be censored at the date of last disease assessment. Progression-free survival will be evaluated using both RECIST 1.1 and immune-related response criteria (irRC), and both sets of results will be reported in each arm. Per RECIST criteria, progression is defined as a >=20% increase in the sum of the longest diameter of the measured lesions, referencing the smallest longest diameter sum, or the appearance of at least one new lesion.
Time Frame: 2 years
Population: 21 subjects were enrolled. One subject withdrew consent before starting treatment and was replaced. A total of 20 patients (10 per each arm) received protocol treatment.
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab + Radiation | Pembrolizumab
Number analyzed (Participants) | 10 | 10
months | 4.5 [2.4 to 20.6] | 6.6 [2.4 to 13.1]

3. Secondary Outcome: Overall Survival (Time From Randomization to Death)
Description: Overall survival is defined as the time from randomization to death or date last known alive. Overall survival will be evaluated using both RECIST 1.1 and immune-related response criteria (irRC), and both sets of results will be reported in each arm. will be evaluated using both RECIST 1.1 and immune-related response criteria (irRC), and both sets of results will be reported in each arm.
Time Frame: 2 years
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab + Radiation | Pembrolizumab
Number analyzed (Participants) | 10 | 10
months | NA [10.1 to NA] — upper limit not reached | 27.2 [22.9 to NA] — upper limit not reached

4. Secondary Outcome: Number of Participants With Complete Response (Absence of Non-irradiated Lesions on Scans)
Description: Complete disappearance of all measurable non-irradiated lesions. All lymph nodes must be non-pathological in size (<10 mm short axis).
Time Frame: 2 years
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Radiation | Pembrolizumab
Number analyzed (Participants) | 10 | 10
Participants | 0 | 0

5. Secondary Outcome: Number of Participants With Partial Response (Tumor Size on Scans)
Description: At least a 30% decrease in the longest diameter valuated using RECIST 1.1.
Time Frame: 2 years
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Radiation | Pembrolizumab
Number analyzed (Participants) | 10 | 10
Participants | 0 | 0

6. Secondary Outcome: Number of Treatment-Emergent Adverse Events
Description: All patients who receive treatment, regardless of eligibility, will be evaluable for toxicity. Toxicity will be graded according to NCI CTCAE, Version 4.0. The proportions of patients with various toxicities will be reported by treatment arm.
Time Frame: 2 years
Population: as for outcome 2
Measure: Number; unit: treatment-emergent adverse events
Arm/Group | Pembrolizumab + Radiation | Pembrolizumab
Number analyzed (Participants) | 10 | 10
treatment-emergent adverse events | 51 | 24

ADVERSE EVENTS:
Time Frame: 2 years
Description: Adverse event evaluation was performed at every protocol visit using the Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v4.0).
Arm/Group | Pembrolizumab + Radiation | Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 1/10 | 1/10
Serious Adverse Events (participants affected / at risk) | 3/10 | 4/10
Other Adverse Events (participants affected / at risk) | 10/10 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab + Radiation (N=10) | Pembrolizumab (N=10)
Hyperthydroidism (Endocrine disorders) | 1 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Elevated ALT (Investigations) | 1 | 0
Elevated AST (Investigations) | 1 | 1
Elevated Alkaline Phosphatase (Investigations) | 1 | 0
Elevated Total Bilirubin (Investigations) | 1 | 0
Aspiration Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Chest Tightness (General disorders) | 0 | 1
Paresthesia (tongue) (Nervous system disorders) | 0 | 1
Confusion (Psychiatric disorders) | 0 | 1
Movement Disorder (tongue and lips) (Nervous system disorders) | 0 | 1
Wound Infection (Infections and infestations) | 0 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab + Radiation (N=10) | Pembrolizumab (N=10)
Alanine Aminotransferase Increased (Investigations) | 2 | 1
Alkaline Phosphatase Increased (Investigations) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Aspartate Aminotransferase Increased (Investigations) | 2 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Chills (General disorders) | 0 | 1
Creatinine Increased (Investigations) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 4 | 0
Dry Mouth (Gastrointestinal disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Endocrine Disorders - Other (Endocrine disorders) | 2 | 0
Fatigue (General disorders) | 4 | 4
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Disorders - Other (Gastrointestinal disorders) | 1 | 0
General Disorders and Administration Site Conditions - Other (General disorders) | 1 | 0
Hepatobiliary Disorders - Other (Hepatobiliary disorders) | 1 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 2
Musculoskeletal and Connective Tissue Disorder - Other (Musculoskeletal and connective tissue disorders) | 2 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Nervous System Disorders - Other (Nervous system disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 1 | 1
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin/Subcutaneous Tissue Disorders - Other (Skin and subcutaneous tissue disorders) | 4 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-28): https://cdn.clinicaltrials.gov/large-docs/19/NCT03087019/Prot_SAP_000.pdf